CLINICAL TRIAL: NCT04293679
Title: An Open Label, Dose Escalation Study to Evaluate the Safety and Efficacy of Intralesional Injection of STP705 in Adult Patients With Cutaneous Squamous Cell Carcinoma in Situ (isSCC)
Brief Title: Open Label, Dose Escalation Study for the Safety and Efficacy of STP705 in Adult Patients With isSCC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRN-705-004
Record Dates: First submitted 2020-02-26; First posted 2020-03-03 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2020-12

CONDITIONS: Bowen's Disease; Cutaneous Squamous Cell Carcinoma in Situ
Keywords: isSCC; Cutaneous Squamous Cell Carcinoma; STP705; Cutaneous Squamous Cell Carcinoma in situ
MeSH Terms: conditions — Bowen's Disease

STUDY DESIGN:
Intervention Model Description: Participants in the first cohort will attend the study center once weekly for an injection of STP705 into the isSCC lesion. The participants will receive injections of STP705 once a week for up to 6 weeks. The clinician will evaluate the tumor for clinical changes and reduction in size at each treatment visit for up to 6 weeks. If during the 6 weeks of treatment there is Complete Clinical Clearance of the tumor, the treatments will end. At the End of Treatment visit, the residual tumor, or former tumor location, will be excised for analysis. In the absence of dose limiting toxicities (DLT), the subsequent cohorts will receive increasing doses of STP705, following the same schedule of administration as the first cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A: STP705 10 μg dose (Experimental): Cohort A: STP705 10 μg dose, intradermal injection, given once a week for up to 6 weeks
  Interventions: Drug: STP705
- Cohort B: STP705 20 μg dose (Experimental): Cohort B: STP705 20 μg dose, intradermal injection, given once a week for up to 6 weeks
  Interventions: Drug: STP705
- Cohort C: STP705 30 μg dose (Experimental): Cohort C: STP705 30 μg dose, intradermal injection, given once a week for up to 6 weeks
  Interventions: Drug: STP705
- Cohort D: STP705 60 μg dose (Experimental): Cohort D: STP705 60 μg dose, intradermal injection, given once a week for up to 6 weeks
  Interventions: Drug: STP705
- Cohort E: STP705 120 μg dose (Experimental): Cohort E: STP705 120 μg dose, intradermal injection, given once a week for up to 6 weeks
  Interventions: Drug: STP705

INTERVENTIONS:
Drug: STP705 — Investigational Product

SUMMARY:
This is an open label, dose escalation study to evaluate the safety and efficacy of intralesional injection of STP705 in adult patients with Cutaneous Squamous Cell Carcinoma in situ (isSCC, Bowen's disease). The purpose of this trial is to evaluate the safety, tolerability and efficacy of various doses of STP705 administered as Intralesional injection in subjects with isSCC.

Goals:

* To determine the safe and effective recommended dose of STP705 for the treatment of isSCC.
* Analysis of biomarkers common to isSCC formation pathway including TGF-β1 and COX-2.

DETAILED DESCRIPTION:
This open label, dose escalation study is designed to evaluate the safety and efficacy of various doses of STP705 administered as an intralesional injection in subjects with cutaneous in situ squamous cell carcinoma (isSCC).

The primary objective of this study is to evaluate the safety, tolerability, and efficacy of various doses of STP705 administered as an Intralesional injection in subjects with cutaneous squamous cell carcinoma in situ skin cancer (isSCC). This study seeks to establish a safe and effective recommended dose of STP705 for the treatment of isSCC. Expression of biomarkers common to the isSCC formation pathway, including TGF-β1 and COX-2, will be evaluated.

The primary endpoint will be the proportion of participants with histological clearance of treated isSCC lesion at the End of Treatment (EOT). Histological clearance (HC) will be defined as the absence of detectable evidence of isSCC tumor cell nests as determined by central pathology review.

Secondary endpoints will include i) time to histological clearance of treated isSCC lesion over the 6 week treatment period, ii) proportion of participants with complete clinical clearance of treated isSCC lesion based on investigator assessment at the End of Treatment (EOT), iii) time to complete clinical clearance of treated isSCC lesion based on investigator assessment over the 6 week treatment period, and iv) the change in size of the treated isSCC lesion over the 6 week treatment period.

Safety and tolerability will be assessed by the number of incidence of adverse events (AEs) and serious adverse events (SAEs); the incidence of AEs and SAEs leading to discontinuation of trial medication; the incidence and severity of Local Skin Response (LSR); hypopigmentation and hyperpigmentation following treatment; and the tolerability of repeated Intralesional administration of STP705 as assessed by investigator-evaluation of injection site reactions for all patients and within each cohort.

In addition, safety measures will include clinically relevant changes or new abnormal findings in laboratory values, vital signs, electrocardiograms (ECGs), and physical examination variables.

25 adult patients are planned to be enrolled in the study. They will be divided equally among 5 cohorts (10, 20, 30, 60 and 120 μg dose levels) of 5 subjects each. Enrollment of the first two subjects in each dosing cohort will be staggered by at least 48 hours. Participants in the first cohort will attend the study center once weekly for an injection of STP705 into the isSCC lesion. The participants will receive injections of STP705 once a week for up to 6 weeks. The clinician will evaluate the tumor for clinical changes and reduction in size at each treatment visit for up to 6 weeks. If during the 6 weeks of treatment there is complete clinical clearance of the tumor, the treatments will end. At the End of Treatment visit, the residual tumor, or former tumor location will be excised for analysis. In the absence of dose limiting toxicities (DLT), the subsequent cohorts will receive increasing doses of STP705, following the same schedule of administration as the first cohort.

If any of the SAEs or dose limiting toxicities outlined above has occurred, the Data Safety Monitoring Board (DSMB) will conduct independent review of the data and will make a final decision for dose escalation to the next cohort.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female adult ≥ 18 years of age.
* 2. Primary, histologically confirmed trunk or extremity (non-peri-orbital/-anogenital/-facial/-scalp) isSCC lesion suitable for excision with a minimum diameter of 0.5cm and with a maximum diameter of 2.0cm.
* 3. Histological diagnosis made no more than 6 months prior to the screening visit.
* 4. Histological biopsy removed ≤25% of the original area of the target lesion.
* 5. No other dermatological disease in the isSCC target site or surrounding area, which in the opinion of the investigator, could interfere with the study.
* 6. Willing to refrain from using non-approved lotions or creams on the target site and surrounding area during the treatment period.
* 7. Willing to refrain from exposure to excessive direct sunlight or ultraviolet light and to avoid the use of tanning parlors for the duration of the study.
* 8. Laboratory values for the tests (listed in the Study Schedule) within the reference ranges as defined by the central laboratory, or "out of range" test results that is clinically acceptable to the investigator. Acceptable "out of range" values are generally those within 2 standard deviations of the mean or explainable due to concurrent medications or disease processes.
* 9. Ability to follow study instructions and likely to complete all study requirements.
* 10. Written informed consent obtained, including consent for tissue to be examined and stored by the Central Histology Lab.
* 11. Written consent to allow photographs of the target isSCC lesion to be used as part of the study data and documentation.
* 12. For females of childbearing potential, a negative pregnancy test at screening and using an acceptable form of birth control (oral / implant/ injectable/ transdermal contraceptives, intrauterine device, condom, diaphragm, abstinence, or a monogamous relationship with a partner who has had a vasectomy).

Exclusion Criteria:

* 1. Pregnant or lactating.
* 2. Presence of known or suspected systemic cancer.
* 3. Histological evidence of nBCC, sBCC, invasive SCC, or any other non-isSCC tumor in the biopsy specimen.
* 4. Histological evidence of severe squamous metaplasia, infiltrative, desomoplastic or micronodular growth patterns in the biopsy specimen.
* 5. History of recurrence of the target isSCC lesion.
* 6. Prior exposure to STP705.
* 7. Evidence of dermatological disease or confounding skin condition in the treatment area, e.g., BCC, actinic keratosis, rosacea, psoriasis, atopic dermatitis, eczema, xeroderma pigmentosa.
* 8. Concurrent disease or treatment that suppresses the immune system;
* 9. Patients with baseline QTC > 480 msec using Frederica's formula
* 10. Chronic medical condition that in the judgment of the investigator(s) would interfere with the performance of the study or would place the patient at undue risk.
* 11. Known sensitivity to any of the ingredients in the study medication.
* 12. Use of a tanning beds or other excessive or prolonged exposure to ultraviolet light or direct sunlight during the study.
* 13. Treatment with systemic chemotherapeutic agents within the 6 months prior to the screening visit.
* 14. Use of systemic retinoids within the 6 months prior to the screening period.
* 15. Treatment with systemic immunomodulators or immunosuppressants within the 6 months prior to the screening period.
* 16. Use of topical immunomodulators within 2cm of the target isSCC lesion within the 4 weeks prior to the screening period.
* 17. Treatment with the following topical agents within 2cm of the target isSCC lesion within the 4 weeks prior to the screening visit: amino-levulanic acid, 5-fluorouracil, corticosteroids, retinoids, diclofenac, ingenol mebutate, or imiquimod.
* 18. Treatment with liquid nitrogen, surgical excision (excluding diagnostic incisional biopsy) or curettage within 2cm of the target isSCC lesion during the 4 weeks prior to the screening visit.
* 19. Elective surgery within 4 weeks prior to the screening visit, during the study, or 4 weeks after the study period.
* 20. Evidence of current chronic alcohol or drug abuse.
* 21. Current enrollment in an investigational drug or device study or participation in such a study within 4 weeks of the screening visit.
* 22. In the investigator's opinion, evidence of unwillingness, or inability to follow the restrictions and requirements of the protocol and complete the study.
* 23. Taking any investigational product within 1 month of first dose of STP705.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with histological clearance of treated isSCC lesion at the End of Treatment (EOT). | 6 weeks
  Proportion of participants with histological clearance of treated isSCC lesion at the End of Treatment (EOT).
  Histological clearance (HC) will be defined as the absence of detectable evidence of isSCC tumor cell nests as determined by central pathology review.

SECONDARY OUTCOMES:
Time to histological clearance of treated isSCC lesion over the 6 week treatment period. | over the 6 week treatment period
Proportion of participants with complete clinical clearance of treated isSCC lesion based on investigator assessment at the End of Treatment (EOT). | 6 weeks
Time to complete clinical clearance of treated isSCC lesion based on investigator assessment over the 6 week treatment period. | over the 6 week treatment period
Change in size of the treated isSCC lesion over the 6 week treatment period. | over the 6 week treatment period
  Change in size of the treated isSCC lesion over the 6 week treatment period. A base line assessment of lesion size will be made by investigator at T1 (first visit, Day 0). The change in size will be assessed every week until the surgical excision of isSCC at the End of Treatment visit (EOT, Day 42) .

CONTACTS AND LOCATIONS:
Overall Officials: Kush Dhody, MBBS, MS, CCRA, Study Director — Amarex Clinical Research, LLC (Amarex); Brian Berman, MD, PhD, Principal Investigator — Center for Clinical and Cosmetic Research
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kuzbicki L, Brozyna AA. Expression of Cyclooxygenase-2 in Human Epithelial Skin Lesions: A Systematic Review of Immunohistochemical Studies. Appl Immunohistochem Mol Morphol. 2021 Mar 1;29(3):163-174. doi: 10.1097/PAI.0000000000000871. PMID 32889812